CLINICAL TRIAL: NCT03151577
Title: Longitudinal Study on Glaucoma Surgery Using XEN® Gel Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Vision Network (Other)
Responsible Party: Principal Investigator, Dr. Kaweh Mansouri, MD, MPH, Swiss Vision Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-02077
Record Dates: First submitted 2017-04-28; First posted 2017-05-12 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: Intraocular pressure, adverse events, complications, number of medications in mild to moderate glaucoma patients who underwent XEN® Gel Stent implantation were recorded.
  Data were collected in a 2 years follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evolution of IOP after XEN® Gel Stent implantation (Other): To study the efficacy of the XEN® Gel Stent in lowering the IOP.
  Interventions: Procedure: XEN® Gel Stent implantation

INTERVENTIONS:
Procedure: XEN® Gel Stent implantation — Minimally invasive glaucoma surgery (MIGS) which consists of implanting a XEN® Gel Stent in the irido-corneal angle of the eye to drain the aqueous humour in the sub-conjunctival space to lower the IOP.
  Other Names: XEN® Gel Stent, Aquesys

SUMMARY:
To evaluate the safety and efficacy of the XEN® Gel Stent in mild to moderate glaucoma patients undergoing glaucoma surgery.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the XEN® Gel Stent in mild to moderate glaucoma patients undergoing glaucoma surgery.

Follow-up period is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate glaucoma patients
* Have given written informed consent
* Aged 18 years or older of either sex

Exclusion Criteria:

* Patients not able to understand the character of the study
* Participation in other clinical research within the last 4 weeks
* Patients with end-stage glaucoma
* Patients with glaucoma surgery done before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Day 0 (=Baseline=before surgery), after surgery on day 1, day 3, week 1, month 1, month 3, month 6, year 1, year 2
  Change in IOP before and after XEN® Gel Stent implantation

SECONDARY OUTCOMES:
Number of needlings | 2 years
  Number of needlings performed during the follow-up after surgery
Number of antiglaucomatous medications | Day 0 (=Baseline=before surgery), after surgery on day 1, day 3, week 1, month 1, month 3, month 6, year 1, year 2
  Change in number of antiglaucomatous medications before and after the surgery.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillmann K, Bravetti GE, Rao HL, Mermoud A, Mansouri K. Bilateral XEN Stent Implantation: A Long-term Prospective Study of the Difference in Outcomes Between First-operated and Fellow Eyes. J Glaucoma. 2020 Jul;29(7):536-541. doi: 10.1097/IJG.0000000000001520. PMID 32341321
- [Derived] Mansouri K, Gillmann K, Rao HL, Guidotti J, Mermoud A. Prospective Evaluation of XEN Gel Implant in Eyes With Pseudoexfoliative Glaucoma. J Glaucoma. 2018 Oct;27(10):869-873. doi: 10.1097/IJG.0000000000001045. PMID 30095603